CLINICAL TRIAL: NCT07182812
Title: Effects of Blood Flow Restriction Sit-to-Stand Exercises on Lumbar Extensor Muscle Endurance, Balance, and Physiological Parameters in Healthy Young Adults: A Randomized Controlled Trial
Brief Title: Effects of Blood Flow Restriction Exercises on Lumbar Muscle Endurance and Balance in Healthy Young Adults
Acronym: BFR-LUMBEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Guler (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Mehmet Akif Guler, PhD, PT, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1919B012413960; 1919B012413960 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers; Low Back Pain; Postural Balance; Muscle Fatigue; Endurance
Keywords: Blood Flow Restriction Exercise; Sit-to-Stand Exercise; Lumbar Extensor Muscles; Muscle Endurance; Postural Balance; Physiological Parameters (Oxygen Saturation, Heart Rate, Blood Pressure); Young Adults; Randomized Controlled Trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial uses a parallel assignment design. Healthy young adults will be randomly allocated into two groups: (1) an experimental group performing sit-to-stand exercises with blood flow restriction (BFR), and (2) a control group performing the same exercises without BFR. Both groups will follow the intervention for six weeks, with two sessions per week. Pre- and post-intervention assessments will be conducted to compare outcomes between groups.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation. Participants and care providers cannot be blinded due to the nature of the intervention (blood flow restriction vs. no restriction). Randomization will be concealed until outcome data collection is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Exercise Group (Experimental): Participants in this arm will perform sit-to-stand exercises combined with blood flow restriction (BFR) using a pneumatic cuff applied to the thigh. The cuff pressure will be set to 60-80% of the participant's systolic blood pressure. The program will be conducted for 6 weeks, with 2 sessions per week, supervised by a physiotherapist.
  Interventions: Behavioral: Blood Flow Restriction Sit-to-Stand Exercise
- Control Exercise Group (Active Comparator): Participants in this arm will perform the same sit-to-stand exercise protocol as the experimental group, but without blood flow restriction. Sessions will also be supervised twice weekly for 6 weeks, and assessments will be performed before and after the intervention.
  Interventions: Behavioral: Sit-to-Stand Exercise without Blood Flow Restriction

INTERVENTIONS:
Behavioral: Blood Flow Restriction Sit-to-Stand Exercise — Participants perform sit-to-stand (STS) exercises with blood flow restriction applied using a pneumatic cuff placed on the thigh. Cuff pressure is set at 60-80% of the participant's systolic blood pressure. Sessions are supervised by a physiotherapist twice per week for six weeks.
  Arms: Blood Flow Restriction Exercise Group
Behavioral: Sit-to-Stand Exercise without Blood Flow Restriction — Participants perform the same sit-to-stand (STS) exercise protocol as the experimental group, but without blood flow restriction. Sessions are supervised twice weekly for six weeks, and outcomes are assessed before and after the program.
  Arms: Control Exercise Group

SUMMARY:
This study aims to examine the effects of blood flow restriction (BFR) exercises on back muscle endurance and balance in healthy young adults. BFR is a training method that involves applying controlled pressure to the limbs with a cuff while performing simple exercises. It has been shown to improve muscle strength and endurance even at low exercise loads, reducing stress on the joints.

In this study, participants aged 20 to 25 years will be randomly assigned to two groups. One group will perform sit-to-stand (STS) exercises combined with BFR, while the other group will perform the same exercises without BFR. The exercise program will last 6 weeks, with 2 sessions per week.

Before and after the program, participants will be assessed for:

Lumbar extensor muscle endurance (using the Biering-Sørensen test)

Balance performance (using a computerized balance platform)

Physiological responses such as oxygen saturation, heart rate, and blood pressure

The purpose of this research is to determine whether BFR exercises improve spinal muscle endurance and balance more effectively than standard sit-to-stand exercises. The results may provide new insights into the use of BFR training as a safe and practical strategy for improving posture, preventing back problems, and enhancing physical performance in young adults.

DETAILED DESCRIPTION:
Detailed Description:

Low back muscle endurance and postural balance are essential components of physical health, functional capacity, and injury prevention. Weakness or fatigue in lumbar extensor muscles is associated with spinal instability, poor posture, and an increased risk of low back pain. Similarly, reduced balance control may impair daily activities and athletic performance. Sedentary lifestyles and prolonged sitting are known to negatively affect these functions in young adults.

Blood flow restriction (BFR) training is an innovative exercise method in which a cuff is applied to partially restrict blood flow in the exercising limb during low-load resistance or functional exercises. This technique has been shown to enhance muscle strength, hypertrophy, and endurance with relatively low mechanical stress, thereby reducing the potential risks associated with high-intensity training. While BFR has been studied extensively in the context of lower-limb strength training, its effects on spinal musculature and balance performance are not well understood.

The present randomized controlled trial is designed to investigate the effects of BFR applied during sit-to-stand (STS) exercises on lumbar extensor muscle endurance and balance performance in healthy young adults. Participants will be randomly assigned to one of two groups:

BFR Exercise Group: STS exercises performed with BFR applied to the thigh.

Control Group: STS exercises performed without BFR.

The intervention will last six weeks, with two supervised exercise sessions per week. The BFR cuff pressure will be set at 60-80% of the individual's systolic blood pressure and monitored to ensure participant safety.

Assessments will be conducted at baseline and after the six-week training program. The primary outcomes are lumbar extensor endurance, measured with the Biering-Sørensen test, and postural balance, assessed using a computerized balance platform. Secondary outcomes include oxygen saturation, heart rate, and blood pressure responses before and after exercise sessions.

The study hypothesizes that participants in the BFR exercise group will show greater improvements in lumbar muscle endurance and balance compared to the control group. Findings from this trial will help clarify whether BFR-based functional training can be considered a safe and effective method not only for enhancing muscle performance but also for improving postural stability in healthy individuals. This may have future applications in sports performance, preventive strategies for low back disorders, and rehabilitation programs for populations with musculoskeletal impairments.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 25 years
* Healthy, without musculoskeletal disorders
* No chronic neurological or systemic disease
* No regular exercise program in the last 3 months
* Voluntary participation with signed informed consent

Exclusion Criteria:

* History of musculoskeletal disease, injury, or chronic low back pain
* Neurological conditions or regular use of medications affecting balance or cardiovascular function
* Pregnancy
* Participation in regular lumbar or core exercise programs within the last 3 months
* Any symptoms during exercise (e.g., excessive fatigue, dizziness, abnormal blood pressure changes) that may pose health risks
* Withdrawal of consent or inability to comply with study protocol

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Lumbar Extensor Muscle Endurance | Baseline and after 6 weeks of intervention
  Endurance of the lumbar extensor muscles will be assessed using the Biering-Sørensen Test. Participants maintain the upper body in a horizontal position while lying prone with the pelvis stabilized. The test duration (in seconds) until trunk decline >5-10° will be recorded.
Postural Balance Performance | Baseline and after 6 weeks of intervention
  Balance performance will be evaluated using a computerized balance platform (TechnoBody™ Pro-Kin). Both static and dynamic balance parameters will be recorded. Outcome measures include sway area (cm²), sway velocity (cm/s), and postural stability index.

SECONDARY OUTCOMES:
Change in Oxygen Saturation | Baseline and immediately after exercise sessions (pre- and post-intervention at 6 weeks)
  Peripheral oxygen saturation (SpO₂, %) will be measured using a pulse oximeter placed on the finger. Measurements will be taken before and after exercise sessions, and changes from baseline to week 6 will be recorded.
Change in Blood Pressure | Baseline and immediately after exercise sessions (pre- and post-intervention at 6 weeks)
  Systolic and diastolic blood pressure will be measured using a validated digital sphygmomanometer. Measurements will be taken at rest before and after exercise sessions. The change from baseline to week 6 will be compared between groups.
Change in Body Mass Index (BMI) | Baseline and after 6 weeks of intervention
  Body mass index (kg/m²) will be calculated from height and weight measured with a digital body composition analyzer (Tanita device). Changes from baseline to week 6 will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Güler, PhD, PT, Principal Investigator — Selçuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Selçuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be available upon reasonable request from qualified researchers after publication of study results. Data will be shared through secure institutional repositories in compliance with Selçuk University ethical guidelines.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the primary results and will be accessible for a period of 5 years thereafter.
Access Criteria: IPD will be available to qualified researchers affiliated with academic or healthcare institutions upon reasonable request. Requests will be reviewed by the principal investigator and Selçuk University Ethics Committee. Approved researchers will gain access through a secure institutional repository with appropriate data use agreements to ensure participant confidentiality.

REFERENCES:
- [Background] Gogna K. Quality assurance: Hodgkin's disease and beyond. Australas Radiol. 2000 Nov;44(4):367-8. doi: 10.1046/j.1440-1673.2000.00839.x. No abstract available. PMID 11103532
- [Background] Meiners KM, Loudon JK. Dynamic and Static Assessment of Single-Leg Postural Control in Female Soccer Players. J Sport Rehabil. 2020 Feb 1;29(2):174-178. doi: 10.1123/jsr.2018-0072. PMID 30526247
- [Background] Madarame H, Neya M, Ochi E, Nakazato K, Sato Y, Ishii N. Cross-transfer effects of resistance training with blood flow restriction. Med Sci Sports Exerc. 2008 Feb;40(2):258-63. doi: 10.1249/mss.0b013e31815c6d7e. PMID 18202577
- [Background] Lee KH, Chon SC. Enhanced Pain Relief and Muscle Growth in Individuals with Low Back Instability: The Impact of Blood Flow Restriction Exercise during Sit to Stand Movements. Med Sci Monit. 2024 Jan 25;30:e942508. doi: 10.12659/MSM.942508. PMID 38268184
- [Background] Loenneke JP, Wilson JM, Marin PJ, Zourdos MC, Bemben MG. Low intensity blood flow restriction training: a meta-analysis. Eur J Appl Physiol. 2012 May;112(5):1849-59. doi: 10.1007/s00421-011-2167-x. Epub 2011 Sep 16. PMID 21922259
- [Background] Demoulin C, Vanderthommen M, Duysens C, Crielaard JM. Spinal muscle evaluation using the Sorensen test: a critical appraisal of the literature. Joint Bone Spine. 2006 Jan;73(1):43-50. doi: 10.1016/j.jbspin.2004.08.002. PMID 16461206
- [Background] Amano S, Ludin AF, Clift R, Nakazawa M, Law TD, Rush LJ, Manini TM, Thomas JS, Russ DW, Clark BC. Effectiveness of blood flow restricted exercise compared with standard exercise in patients with recurrent low back pain: study protocol for a randomized controlled trial. Trials. 2016 Feb 12;17:81. doi: 10.1186/s13063-016-1214-7. PMID 26867541